CLINICAL TRIAL: NCT06191562
Title: Randomized Clinical Trial of Post-operative Outcomes Following Posterior Versus Anterior Tympanostomy Tube Placement
Brief Title: Posterior Vs. Anterior Tympanostomy Tube Placement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Chi, MD (Other)
Responsible Party: Sponsor-Investigator, David Chi, MD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY22120108
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Otitis Media in Children; Chronic Otitis Media with Effusion; Recurrent Acute Otitis Media
Keywords: Middle ear ventilation; Otitis media
MeSH Terms: conditions — Otitis Media | interventions — Middle Ear Ventilation

STUDY DESIGN:
Intervention Model Description: Experimental, randomized control trial with no placebo
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Posterior Tympanostomy Tube Left (Experimental): Patients in whom the left ear is randomized to receive a tympanostomy tube in the posterior-inferior quadrant (new location).
  Interventions: Device: Tympanostomy tube
- Posterior Tympanostomy Tube Right (Experimental): Patients in whom the right ear is randomized to receive a tympanostomy tube in the posterior-inferior quadrant (new location).
  Interventions: Device: Tympanostomy tube

INTERVENTIONS:
Device: Tympanostomy tube — Participants will receive an ear tube in the usual location (anterior-inferior) in one ear and a new location (posterior-inferior) in the other ear during surgery.
  Other Names: Myringotomy with tubes; pressure equalization tubes; ventilation tubes

SUMMARY:
The goal of this randomized clinical trial is to compare the results of ear tube placement in two different parts of the ear drum. The ear drum can be divided into four parts (called quadrants). Ear tubes are usually placed in one section of the ear drum, called the anterior-inferior quadrant. However, tubes can also be placed in another section, called the posterior-inferior quadrant. Ear tubes usually fall out of the ear drum on their own. In most patients, the hole in the ear drum where the tube used to be closes on its own. Sometimes (in about 2% of patients), the hole does not close on its own and might need surgery. We want to study ear tube placement in the posterior-inferior quadrant because surgery to repair a hole in the eardrum is easier in this location.

For this study, children will receive an ear tube in the usual location (anterior-inferior quadrant) in one ear and the new location (posterior-inferior quadrant) in the other ear. Researchers will determine which ear has the new location using random assignment (like flipping a coin). Researchers will collect information about hearing tests, whether there is ear drainage (otorrhea), if the tube is blocked (occluded), and how the ear drum looks for up to 37 months after tube placement. Participants will answer study questions at 2-12 weeks and 6, 12, 18, 24, 30, and 36 months after surgery. These questions will ask about whether tubes have fallen out of the ear drum, whether there is a hole in the ear drum, whether there has been drainage from the ear or other ear symptoms, and whether there have been any visits to the doctor for ear problems.

Researchers will use this information to compare ears with anterior-inferior tube placement and ears with posterior-inferior tube placement to see if there are differences in common complications following tube placement.

DETAILED DESCRIPTION:
The tympanic membrane can be divided into quadrants: posterior superior, anterior superior, posterior inferior, and anterior inferior. Traditional training dictates that tympanostomy tubes should be placed in the anterior-inferior quadrant, with the thought that this would lead to longer indwelling time in the tympanic membrane, avoidance of damage to the ossicular chain, and prevention of hearing loss due to residual perforation over the round window following tympanostomy tube extrusion. However, more recent work has challenged these assumptions. Notably, there is a 2-16% risk of chronic perforation following tympanostomy tube extrusion, with a proposed annual incidence of more than 40,000 post-tympanostomy tube perforations in the United States each year. While perforations in the posterior tympanic membrane can often be repaired using transcanal approaches, anterior perforations are more likely to require more invasive postauricular or endoaural approaches or canalplasty. To our knowledge, there are no studies reporting outcomes following tympanostomy tube placement in the posterior-inferior quadrant. If this study demonstrates no difference in hearing, tube indwelling time, and sequelae following posterior-inferior placement compared with anterior-inferior, it would allow otolaryngologists greater flexibility to consider patient characteristics such as factors placing them at increased risk for perforation or anatomy of the auditory canal when selecting the section of tympanic membrane in which to place tubes.

Upon completion of screening, patients will be randomized using a random number generator in order to have an equal distribution of left and right ears with tympanostomy tubes placed in the anterior and posterior quadrants. Consented patients will receive an ear tube in the usual location (anterior-inferior) in one ear and a new location (posterior-inferior) in the other ear during surgery. Follow-up will include standard-of-care post-operative visits and may be completed at 2-12 weeks and 5-7 months. Clinicians will examine the child's ears and determine whether otorrhea and occlusion are present. During the visit, audiologists may conduct standard of care ear-specific pure tone average, air-bone gap, and sound field audiometry. At these follow-up visits, otolaryngology providers will complete a form describing the status of the tympanic membrane. This will add <1 minute to the visit. Caregivers will also complete a form asking about the status of their child's tympanostomy tubes and any ear problems their child has experienced since surgery. This will take <5 minutes to complete. Results of audiology testing will be collected from the electronic medical record. Additional follow-up will include administration of the caregiver questions via phone, mail, or REDCap email at 12, 18, 24, 30, and 36 months. If the child has other follow-up clinic visits prior to 37 months post-surgery, the provider form will be completed again during these visits. Further research activities will include viewing medical charts of the included subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 6 months -14 years
2. Bilateral tympanostomy tube placement
3. First tympanostomy tubes placement
4. Indication for tympanostomy tube placement is otitis media

Exclusion Criteria:

1. Undergoing tympanostomy tube placement for indication other than otitis media
2. Receiving tubes other than Armstrong grommet.
3. Genetic disorder that impacts the craniofacial structure, immune system, or mucosal secretions such as Downs syndrome, Stickler syndrome, Treacher Collins syndrome, other genetic disorder associated with craniofacial anomalies, Severe Combined Immunodeficiency disorder, Cystic Fibrosis, or Primary Ciliary Dyskinesia
4. Patients with craniofacial abnormalities other than plagiocephaly or submucous cleft palate (SMCP)
5. Caregivers who cannot speak, read, or write in English proficiently
6. Prior or current otologic surgery other than tympanostomy tube placement
7. On systemic corticosteroids at the time of enrollment
8. Immunodeficiency (acquired or congenital)
9. Current retraction, cholesteatoma, or middle ear mass
10. Atresia
11. Sensorineural hearing loss
12. Known ossicular chain anomaly

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 386 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Perforation | Within 36 months +/- 30 days following tympanostomy tube placement
  Percentage of ears with persistent (>3 month) perforation of the tympanic membrane

SECONDARY OUTCOMES:
Parent-reported otorrhea at 2-12 weeks | 2-12 weeks following tympanostomy tube placement
  Percentage of ears with ear drainage most days (67-100%), many days (33-67%), some days (1-33%) or no days (0)
Parent-reported otorrhea at 6 months | 6 months±30 days following tympanostomy tube placement
  Percentage of ears with ear drainage most days (67-100%), many days (33-67%), some days (1-33%) or no days (0)
Provider-observed tube occlusion at 2-12 weeks | 2-12 weeks following tympanostomy tube placement
  Percentage of ears with tubes occluded
Provider-observed tube occlusion at 6 months | 6 months±30 days following tympanostomy tube placement
  Percentage of ears with tubes occluded
Provider-observed tympanostomy tubes in place and patent at 2-12 weeks | 2-12 weeks following tympanostomy tube placement
  Percentage of ears with tympanostomy tubes in place and patent
Provider-observed tympanostomy tubes in place and patent at 6 months | 6 months±30 days following tympanostomy tube placement
  Percentage of ears with tympanostomy tubes in place and patent
Retained tubes requiring surgical intervention | Within 36 months +/- 30 days following tympanostomy tube placement
  Percentage of ears requiring surgical tympanostomy tube removal
Perforation requiring surgical intervention | Within 36 months +/- 30 days following tympanostomy tube placement
  Percentage of ears with surgical repair of perforation
Atrophy or retraction at tube site | Within 36 months +/- 30 days following tympanostomy tube placement
  Percentage of ears with atrophy or retraction at tube site
Cholesteatoma | Within 36 months +/- 30 days following tympanostomy tube placement
  Percentage of ears with cholesteatoma
Hearing loss | Within 36 months +/- 30 days following tympanostomy tube placement
  Percentage of ears with pure tone average >20 dB or absent otoacoustic emissions
Tube indwelling time before extrusion | Within 36 months +/- 30 days following tympanostomy tube placement
  Months from tympanostomy tube placement to extrusion estimated from parent-report and provider observations
Ability to see through lumen and assess tube patency at 2-12 weeks | 2-12 weeks following tympanostomy tube placement
  Percentage of ears in which the otolaryngology provider is able to see through lumen and assess tube patency
Ability to see through lumen and assess tube patency at 6 months | 6 months±30 days following tympanostomy tube placement
  Percentage of ears in which the otolaryngology provider is able to see through lumen and assess tube patency

OTHER OUTCOMES:
Parent-reported otorrhea at 12 months | 12 months±30 days following tympanostomy tube placement
  Percentage of ears with ear drainage most days (67-100%), many days (33-67%), some days (1-33%) or no days (0)
Parent-reported otorrhea at 18 months | 18 months±30 days following tympanostomy tube placement
  Percentage of ears with ear drainage most days (67-100%), many days (33-67%), some days (1-33%) or no days (0)
Parent-reported otorrhea at 24 months | 24 months±30 days following tympanostomy tube placement
  Percentage of ears with ear drainage most days (67-100%), many days (33-67%), some days (1-33%) or no days (0)
Parent-reported otorrhea at 30 months | 30 months±30 days following tympanostomy tube placement
  Percentage of ears with ear drainage most days (67-100%), many days (33-67%), some days (1-33%) or no days (0)
Parent-reported otorrhea at 36 months | 36 months±30 days following tympanostomy tube placement
  Percentage of ears with ear drainage most days (67-100%), many days (33-67%), some days (1-33%) or no days (0)
Parent-reported blockage of tube lumen at 2-12 weeks | 2-12 weeks following tympanostomy tube placement
  Percentage of ears clogged/blocked
Parent-reported blockage of tube lumen at 6 months | 6 months±30 days following tympanostomy tube placement
  Percentage of ears clogged/blocked
Parent-reported blockage of tube lumen at 12 months | 12 months±30 days following tympanostomy tube placement
  Percentage of ears clogged/blocked
Parent-reported blockage of tube lumen at 18 months | 18 months±30 days following tympanostomy tube placement
  Percentage of ears clogged/blocked
Parent-reported blockage of tube lumen at 24 months | 24 months±30 days following tympanostomy tube placement
  Percentage of ears clogged/blocked
Parent-reported blockage of tube lumen at 30 months | 30 months±30 days following tympanostomy tube placement
  Percentage of ears clogged/blocked
Parent-reported blockage of tube lumen at 36 months | 36 months±30 days following tympanostomy tube placement
  Percentage of ears clogged/blocked
Provider-observed otorrhea at 2-12 weeks | 2-12 weeks following tympanostomy tube placement
  Percentage of ears with otorrhea observed by provider
Provider-observed otorrhea at 6 months | 6 months±30 days following tympanostomy tube placement
  Percentage of ears with otorrhea observed by provider
Provider-observed otorrhea at 12 months | 12 months±30 days following tympanostomy tube placement
  Percentage of ears with otorrhea observed by provider
Provider-observed otorrhea at 18 months | 18 months±30 days following tympanostomy tube placement
  Percentage of ears with otorrhea observed by provider
Provider-observed otorrhea at 24 months | 24 months±30 days following tympanostomy tube placement
  Percentage of ears with otorrhea observed by provider
Provider-observed otorrhea at 30 months | 30 months±30 days following tympanostomy tube placement
  Percentage of ears with otorrhea observed by provider
Provider-observed otorrhea at 36 months | 36 months±30 days following tympanostomy tube placement
  Percentage of ears with otorrhea observed by provider
Provider-observed tube occlusion at 12 months | 12 months±30 days following tympanostomy tube placement
  Percentage of ears with tubes occluded
Provider-observed tube occlusion at 18 months | 18 months±30 days following tympanostomy tube placement
  Percentage of ears with tubes occluded
Provider-observed tube occlusion at 24 months | 24 months±30 days following tympanostomy tube placement
  Percentage of ears with tubes occluded
Provider-observed tube occlusion at 30 months | 30 months±30 days following tympanostomy tube placement
  Percentage of ears with tubes occluded
Provider-observed tube occlusion at 36 months | 36 months±30 days following tympanostomy tube placement
  Percentage of ears with tubes occluded
Provider-observed tympanostomy tubes in place and patent at 12 months | 12 months±30 days following tympanostomy tube placement
  Percentage of ears with tympanostomy tubes in place and patent
Provider-observed tympanostomy tubes in place and patent at 18 months | 18 months±30 days following tympanostomy tube placement
  Percentage of ears with tympanostomy tubes in place and patent
Provider-observed tympanostomy tubes in place and patent at 24 months | 24 months±30 days following tympanostomy tube placement
  Percentage of ears with tympanostomy tubes in place and patent
Provider-observed tympanostomy tubes in place and patent at 30 months | 30 months±30 days following tympanostomy tube placement
  Percentage of ears with tympanostomy tubes in place and patent
Provider-observed tympanostomy tubes in place and patent at 36 months | 36 months±30 days following tympanostomy tube placement
  Percentage of ears with tympanostomy tubes in place and patent
Ability to see through lumen and assess tube patency at 12 months | 12 months±30 days following tympanostomy tube placement
  Percentage of ears in which the otolaryngology provider is able to see through lumen and assess tube patency
Ability to see through lumen and assess tube patency at 18 months | 18 months±30 days following tympanostomy tube placement
  Percentage of ears in which the otolaryngology provider is able to see through lumen and assess tube patency
Ability to see through lumen and assess tube patency at 24 months | 24 months±30 days following tympanostomy tube placement
  Percentage of ears in which the otolaryngology provider is able to see through lumen and assess tube patency
Ability to see through lumen and assess tube patency at 30 months | 30 months±30 days following tympanostomy tube placement
  Percentage of ears in which the otolaryngology provider is able to see through lumen and assess tube patency
Ability to see through lumen and assess tube patency at 36 months | 36 months±30 days following tympanostomy tube placement
  Percentage of ears in which the otolaryngology provider is able to see through lumen and assess tube patency
Ear-specific pure tone average | Within 36 months +/- 30 days following tympanostomy tube placement
  Highest (worst) pure tone average of 500 Hz, 1000 Hz, 2000 Hz, and 3000 Hz in decibels
Ear-specific speech-response threshold | 36 months±30 days following tympanostomy tube placement
  Highest (worst) speech-response threshold in decibels
Ear-specific speech-awareness threshold | Within 36 months +/- 30 days following tympanostomy tube placement
  Highest (worst) speech-awareness threshold in decibels

CONTACTS AND LOCATIONS:
Overall Officials: David H Chi, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh North, Sewickley, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in a publication may be shared, after de-identification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 1 year after publication of summary data. Ending 5 years after publication.
Access Criteria: IPD will be shared with researchers who provide a methodologically sound proposal. IPD to be shared will include that necessary to achieve the aims in the approved proposal. Proposals should be directed to shafferad@upmc.edu. To gain access, data requestors will need to sign data access agreement.

REFERENCES:
- [Background] ALBERTI PW. EPITHELIAL MIGRATION ON THE TYMPANIC MEMBRANE. J Laryngol Otol. 1964 Sep;78:808-30. doi: 10.1017/s0022215100062800. No abstract available. PMID 14205963
- [Background] O'Donoghue GM. The kinetics of epithelial cells in relation to ventilating tubes. Acta Otolaryngol. 1984 Jul-Aug;98(1-2):105-9. doi: 10.3109/00016488409107541. PMID 6380208
- [Background] Gibb AG, Mackenzie IJ. The extrusion rate of grommets. Otolaryngol Head Neck Surg. 1985 Dec;93(6):695-9. doi: 10.1177/019459988509300601. PMID 3937089
- [Background] Kivekas I, Poe D. Is there an optimal location for tympanostomy tube placement? Laryngoscope. 2015 Jul;125(7):1513-4. doi: 10.1002/lary.25127. Epub 2015 Jan 13. No abstract available. PMID 25582620
- [Background] Mehta RP, Rosowski JJ, Voss SE, O'Neil E, Merchant SN. Determinants of hearing loss in perforations of the tympanic membrane. Otol Neurotol. 2006 Feb;27(2):136-43. doi: 10.1097/01.mao.0000176177.17636.53. PMID 16436981
- [Background] Stinson WD. Reparative processes in the membrana tympani: some interested manifestations. Arch Otolaryngol. 1936; 24(5): 600-605. doi:10.1001/archotol.1936.00640050613006.